CLINICAL TRIAL: NCT04900142
Title: Micropulsed Laser Trabeculoplasty: a Randomized Double Blinded Clinical Trial Using Different Parameters
Brief Title: Micropulsed Laser Trabeculoplasty Using Different Parameters
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Modena and Reggio Emilia (Other)
Responsible Party: Principal Investigator, Gian Maria Cavallini, Associate Professor, University of Modena and Reggio Emilia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1152/2019/DISP/AOUMO
Record Dates: First submitted 2020-12-19; First posted 2021-05-25 (Actual); Last update posted 2021-05-25 (Actual); Status verified 2021-05

CONDITIONS: Glaucoma, Open-Angle
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1500 mW (Experimental): 1500 mW of Power
  Interventions: Procedure: Micropulsed laser trabeculoplasty
- 1000 mW (Active Comparator): Standard treatment, 1000 mW
  Interventions: Procedure: Micropulsed laser trabeculoplasty

INTERVENTIONS:
Procedure: Micropulsed laser trabeculoplasty — Trabeculoplasty

SUMMARY:
This randomized, double blinded, clinical trial compares two different parameters setting of micropulsed laser trabeculoplasty for open angle glaucoma. Group one is treated with 1500 mW of Power, Group two with 1000 mW. The other settings (300 micron of diameter, 300 ms of duration, 15% duty cycle) are the same for both groups, and the laser is applied for 360°.

The main outcome is to evaluate the IOP (IntraOcular Pressure) lowering effects of both treatments and the safety on the corneal endothelium.

DETAILED DESCRIPTION:
This study is a randomized, double blinded, clinical trial. Eligibility criteria are: primary open angle glaucoma, pigmentary glaucoma and pseudoexfoliation glaucoma.

Exclusion criteria are: secondary glaucoma, previous glaucoma surgery (not including cataract surgery as a glaucoma surgery), uncooperative patients, corneal endothelial diseases (such as Fuchs dystrophy or cornea guttata) and severely decompensated glaucoma.

Both eyes of the patient are treated: each eye is allocated in a group using the closed envelopes method. Both the patient and the surgeon who performs the post laser examinations are not aware of the group allocation.

The exams required before the trabeculoplasty are: best corrected visual acuity, IOP measurement, specular microscopy with corneal central thickness.

The IOP is measured an hour after MLT (micropulsed laser trabeculoplasty), then on day one, at one month, at three months and six months. Best corrected visual acuity and specular microscopy are repeated at three months.

Expected outcomes: to compare the IOP lowering effects between group one and two and to assess the safety of the procedure on the corneal endothelium.

Secondary outcomes: decrease the number of glaucoma medications applied by the patients.

ELIGIBILITY:
Inclusion Criteria:

* Primary open angle glaucoma
* Pigmentary glaucoma
* Pseudoexfoliative glaucoma

Exclusion Criteria:

* Secondary glaucoma
* Previous glaucoma surgery
* Severely decompensated glaucoma
* Corneal endothelial disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-03-20 (Actual); Primary Completion 2022-03-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
IOP lowering effect | Up to six months
  Using a tonometer, we will evaluate the difference in intraocular pressure between baseline and after the treatment. The values will be expressed in mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Mastropasqua Rodolfo, MD, Professor, Study Director — Policlinico di Modena
Locations (1):
- Policlinico di Modena, Modena, Italy